CLINICAL TRIAL: NCT05331690
Title: A Randomized Clinical Three-arm Trial Comparing Inflammation and Cystoid Macular Edema for the Medication Regimens Preoperative and Postoperative Topical NSAIDs to Only Postoperative Topical NSAIDs to Postoperative Topical NSAIDs and Steroids in Patients Undergoing Cataract Surgery (Pre-CIN).
Brief Title: Cataract Surgery and Inflammation - the Role for Preoperative NSAIDs (Pre-CIN)
Acronym: pre-CIN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Olav Kristianslund, Principal investigator, Head of section / Senior consultant MD PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 93944; 2020-003407-34 (EudraCT Number)
Record Dates: First submitted 2022-04-09; First posted 2022-04-18 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Cataract Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 NSAIDs pre (Active Comparator): Topical nepafenac (Nevanac) 3 mg/ml started 1 day before surgery
  Interventions: Drug: Nepafenac Ophthalmic
- Group 2 NSAIDs post (Active Comparator): Topical nepafenac (Nevanac) 3 mg/ml started the day after surgery
  Interventions: Drug: Nepafenac Ophthalmic
- Group 3 NSAIDs and steroids (Active Comparator): Topical nepafenac (Nevanac) 3 mg/ml + topical dexamethasone (Spersadex) started the day after surgery
  Interventions: Drug: Nepafenac Ophthalmic; Drug: Dexamethasone Ophthalmic

INTERVENTIONS:
Drug: Nepafenac Ophthalmic — Topical nepafenac (Nevanac) 3 mg/ml starter the day before surgery
  Arms: Group 1 NSAIDs pre
Drug: Nepafenac Ophthalmic — Topical nepafenac (Nevanac) 3 mg/ml started the day after surgery
  Arms: Group 2 NSAIDs post; Group 3 NSAIDs and steroids
Drug: Dexamethasone Ophthalmic — Topical dexamethasone 1 mg/ml (Spersadex) started the day after surgery
  Arms: Group 3 NSAIDs and steroids

SUMMARY:
The pre-CIN trial is a randomized clinical three-arm trial comparing inflammation and cystoid macular edema for the medication regimens preoperative and postoperative topical NSAIDs to only postoperative topical NSAIDs to postoperative topical NSAIDs and steroids in patients undergoing cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years and older at the time of the signing of the informed consent. There is no upper age limit.
* Scheduled for standard phacoemulsification cataract surgery (group 1 - 3)
* Scheduled for combined phacoemulsification cataract surgery and MIGS stent (group 4)
* Ability to cooperate fairly well during the examinations
* Willing to participate in the study and capable of giving informed consent, which includes compliance with the requirements and restrictions in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Contraindications for use of any medication (as listed in the approved SPC, e.g. allergy, pregnancy, breastfeeding)
* Pregnancy
* Diabetes
* Mature cataract
* Active or chronic uveitis with recommendation for steroid treatment
* Previous trabeculectomy
* Other ophthalmological conditions and/or complicating factors requiring steroid treatment (group 1 - 3)
* Cornea pathology requiring specific medication regimens (e.g. herpes pathology, previous corneal transplantation)

Patients with complications or other complicating factors during surgery that causes the surgeon to demand both NSAIDs and steroid treatment will be excluded from the main analysis. These patients will be followed postoperatively as part of the study and included in additional analyses (for example as part of an intention to treat analysis).

For patients scheduled for cataract surgery in both eyes, only the first operated eye will be included, however, both eyes will be examined.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Central macular thickness after 6 weeks | 6 weeks after surgery
  Measure central macular thickness (in um) on optical coherence tomography (OCT)
Cystoid macular edema (CME) after 6 weeks | 6 weeks after surgery
  Determine if the patient has CME based on evaluation of macular cysts on optical coherence tomography (OCT)

SECONDARY OUTCOMES:
Intraocular inflammation | Preoperatively, and 1 week, 6 weeks, 6 months after surgery
  Measured by laser flare meter
Visual outcome | Preoperatively, and 1 week, 6 weeks, 6 months after surgery
  Measure uncorrected and corrected distance visual acuity using visual acuity chart
Intraocular pressure | Preoperatively, and 1 week, 6 weeks, 6 months after surgery
  Measured by tonometry
Central macular thickness (CMT) | Preoperatively, 1 week, and 6 months after surgery
  Measure CMT (in um) on optical coherence tomography (OCT)
Cystoid macular edema (CME) | Preoperatively, 1 week, and 6 months after surgery
  Determine if the patient has CME based on evaluation of macular cysts on optical coherence tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Olav Kristianslund, MD PhD, Principal Investigator — Department of Ophthalmology, Oslo University Hospital
Locations (1):
- Department of Ophthalmology, Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided